CLINICAL TRIAL: NCT00874029
Title: Evaluation of the Halt System for Laparoscopic Treatment of Symptomatic Uterine Fibroids With Radiofrequency Ablation
Brief Title: Laparoscopic Radiofrequency Ablation (RFA) of Symptomatic Uterine Fibroids
Acronym: Halt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acessa Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00-0004
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Uterine Fibroids; Uterine Myomas
Keywords: Uterine Fibroids; Myomas
MeSH Terms: conditions — Leiomyoma; Myoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Halt Procedure (Experimental): In this single-arm study, subjects who have symptomatic uterine fibroids will have the Halt Procedure in which intra-abdominal ultrasound will guide RF ablation of uterine fibroids using the Halt System.
  Interventions: Device: Halt Procedure

INTERVENTIONS:
Device: Halt Procedure — The Halt 2000 Electrosurgical Radiofrequency Ablation System is indicated for use in percutaneous, laparoscopic and intraoperative, coagulation and ablation of soft tissue.
  Other Names: Halt; Halt2000; The Halt System; The Halt 2000 System

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of radiofrequency ablation (RFA) using the Halt System for the treatment of patients with symptomatic uterine fibroids.

DETAILED DESCRIPTION:
In this single-arm study, subjects who have symptomatic uterine fibroids will have laparoscopic surgery in which intra-abdominal ultrasound will guide RF ablation of uterine fibroids using the Halt System.

ELIGIBILITY:
Inclusion Criteria:

* Are premenopausal and ≥ 25 years old
* Have symptomatic uterine fibroids
* Have a uterine gestational size ≤14 weeks as determined by pelvic exam
* Have ≤ 6 (six) treatable fibroids in whom no single fibroid exceeds 7 cm in any diameter as measured by ultrasound or magnetic resonance imaging (MRI). Only Fibroids greater than 1cm in diameter should be treated in this study
* Have a total uterine fibroid volume that does not exceed 300cc on ultrasound or contrast-enhanced MRI evaluation
* Have clinical menorrhagia as indicated by menstrual blood loss of ≥160 mL to 500 ml during one baseline cycle or two baseline cycles within three months prior to treatment
* Have a history of at least 3 months of menorrhagia within the last six months
* Desire uterine preservation
* Do not desire current or future childbearing
* Have a normal coagulation profile international normalized ratio (INR), Platelets, Prothrombin Time, and Partial Thromboplastin Time (PTT)
* Have had a normal Pap smear within the past 12 months
* Are practicing non-hormonal or stable hormonal contraception
* If the woman is not currently taking any hormonal contraceptives, has been off all hormonal contraceptives for a minimum of three months prior to study enrollment, and agrees to continue without change in regimen through the 12 months of follow-up OR
* If the woman is currently taking hormonal contraceptives, has taken hormonal contraceptives for a minimum of three months prior to study enrollment, and agrees to continue without change in regimen through 12 months of follow up.**

  **Note: Hormonal contraceptive use must be terminated 30 days prior to treatment but should be resumed post-operatively within 60 days post treatment as instructed by the Investigator.
* Are willing and able to comply with all study tests, procedures, and assessment tools
* Are willing and able to return for all required follow up visits following study enrollment
* Must pass a pre-operative health exam (ASA I-III)
* Are capable of providing informed consent

Exclusion Criteria:

* Have contraindications for laparoscopic surgery and/or general anesthesia. (Contraindications include anemia, defined as a hemoglobin level under 10 or hematocrit level less than 30.)
* Have had prior pelvic surgery (with the exception of C-section, tubal ligation, or diagnostic laparoscopy), or are known to have significant intra-abdominal adhesions (defined as adhesions that would require extensive dissection to mobilize and view all surfaces of the uterus)
* Have previously undergone endometrial ablation, uterine artery embolization, or uterine artery ligation, or any other uterine-preserving technique for reduction of menstrual bleeding (with the exception of hysteroscopic myomectomy > 1 year ago)
* Patients requiring elective concomitant procedures
* Have contraindications for magnetic resonance imaging (MRI)
* Desire current or future childbearing
* Are pregnant or lactating
* Have taken any Gonadotropin-releasing hormone (GnRh) agonist within three months prior to the screening procedures
* Have an implanted intrauterine or fallopian tube device for contraception that cannot or will not be removed one month prior to treatment
* Have dysfunctional uterine bleeding or bleeding between periods
* Have chronic pelvic pain not due to uterine fibroids
* Have known or suspected endometriosis
* Have known or suspected adenomyosis based on Ultrasound or MRI findings
* Have active or history of pelvic inflammatory disease
* Have a history of or evidence of gynecologic malignancy or pre-malignancy within the past five years
* Have had pelvic radiation
* Have a non-uterine pelvic mass
* Have a cervical myoma
* Have one or more pedunculated subserosal fibroids or "type zero" (completely intracavitary) submucous fibroids
* Are peri-menopausal (defined as women 40 years of age or older with Follicular Stimulating Hormone level of ≥ 25 International Units (IU) or menopausal
* Are unable to give informed consent
* In the medical judgment of the investigator should not participate in the study

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hinckley, MD, Principal Investigator — Reproductive Science Center; Micah Harris, MD, Principal Investigator — Women's Health Research; Erika Banks, MD, Principal Investigator — Montefiore Medical Center; Karen R Abbott, MD, Principal Investigator — Athena Gynecology Medical Group; Jay Berman, MD, Principal Investigator — Wayne State University; Jose G Garza Leal, MD, Principal Investigator — Hospital Universitario Dr. Jose Eleuterio Gonzalez; David Levine, MD, Principal Investigator — St. Johns' Mercy Medical Center; Rodolfo Robles Pemueller, MD, Principal Investigator — Universidad Francisco Marroquín; Jennifer Israel, MD, Principal Investigator — University of Southern California; Richard S Guido, MD, Principal Investigator — Magee-Women's Hospital; James Macer, MD, Principal Investigator — Pasadena Premier Women's Health
Locations (11):
- United States (9):
  - Women's Health Research, Phoenix, Arizona
  - USC Medical Center, Los Angeles, California
  - Pasadena Premier Women's Health, Pasadena, California
  - Reproductive Science Center, San Ramon, California
  - Wayne State University, Detroit, Michigan
  - St. Luke's Hospital, Chesterfield, Missouri
  - Athena Gynecology Medical Group, Reno, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
- Hospital Universitario Esperanza, Guatemala City, Departamento de Guatemala, Guatemala
- Hospital Universitario Dr. Jose Eleuterio Gonzalez de la Universidad Autonoma de Nuevo Leon. Facultad de Medicina, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Result] Chudnoff SG, Berman JM, Levine DJ, Harris M, Guido RS, Banks E. Outpatient procedure for the treatment and relief of symptomatic uterine myomas. Obstet Gynecol. 2013 May;121(5):1075-1082. doi: 10.1097/AOG.0b013e31828b7962. PMID 23635746
- [Result] Robles R, Aguirre VA, Argueta AI, Guerrero MR. Laparoscopic radiofrequency volumetric thermal ablation of uterine myomas with 12 months of follow-up. Int J Gynaecol Obstet. 2013 Jan;120(1):65-9. doi: 10.1016/j.ijgo.2012.07.023. Epub 2012 Oct 14. PMID 23073229
- [Result] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Lee BB. Laparoscopic ultrasound-guided radiofrequency volumetric thermal ablation of symptomatic uterine leiomyomas: feasibility study using the Halt 2000 Ablation System. J Minim Invasive Gynecol. 2011 May-Jun;18(3):364-71. doi: 10.1016/j.jmig.2011.02.006. PMID 21545960
- [Result] Guido RS, Macer JA, Abbott K, Falls JL, Tilley IB, Chudnoff SG. Radiofrequency volumetric thermal ablation of fibroids: a prospective, clinical analysis of two years' outcome from the Halt trial. Health Qual Life Outcomes. 2013 Aug 13;11:139. doi: 10.1186/1477-7525-11-139. PMID 23941588
- [Derived] Levine DJ, Berman JM, Harris M, Chudnoff SG, Whaley FS, Palmer SL. Sensitivity of myoma imaging using laparoscopic ultrasound compared with magnetic resonance imaging and transvaginal ultrasound. J Minim Invasive Gynecol. 2013 Nov-Dec;20(6):770-4. doi: 10.1016/j.jmig.2013.04.015. Epub 2013 Sep 8. PMID 24021910
- [Derived] Galen DI, Isaacson KB, Lee BB. Does menstrual bleeding decrease after ablation of intramural myomas? A retrospective study. J Minim Invasive Gynecol. 2013 Nov-Dec;20(6):830-5. doi: 10.1016/j.jmig.2013.05.007. Epub 2013 Sep 7. PMID 24018147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2009 with enrollment of the last patient in February 2011. All subjects were enrolled at nine clinical sites throughout the United States and two clinical sites in Latin America.
Pre-assignment Details: Subjects were excluded for the following: radiologic evidence by MRI of adenomyosis (n = 127), pedunculated subserosal or intracavitary myomas (n = 43), a history of pelvic malignancy, cervical dysplasia, a prior procedure to treat or remove myomas (n = 22), and contraindications to anesthesia or abdominal surgery (n = 12).
Period: Overall Study
Arm/Group | Halt Procedure
Started | 137
Completed | 116
Not Completed | 21
Not completed — Withdrawal by Subject | 10
Not completed — Pregnancy | 4
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: Subjects who met the initial inclusion exclusion criteria were enrolled and treated. Two subjects were later found to have baseline bleeding volumes outside of the protocol inclusion limits. All 137 Subjects comprised the Safety Set. The Full Analysis Set excluded the two subjects that did not meet the baseline bleeding criteria.
Groups:
- Halt Medical Acessa Procedure: In this single-arm study, subjects who have symptomatic uterine fibroids had the Acessa Procedure using the Halt Medical Proprietary Acessa System. The Acessa System delivers monopolar radiofrequency energy to tissue through a disposable electrosurgical radiofrequency (RF) Handpiece. The Generator provides sinusoidally-varying voltage at 460 kilohertz (kHz) to drive a current through the tissue to be ablated. The current delivered through the Handpiece causes controlled, local heating, resulting in targeted tissue destruction. The heat produced then disperses by conduction. During these controlled ablations, the Generator produces an alternating current which flows between the Handpiece and the dispersive electrode pads, through the body of the patient. These components, coupled with the visualization capabilities of laparoscopic ultrasound, enable the surgeon to accurately identify the patient's uterine fibroids and treat all of her fibroids, and just the fibroids.
Arm/Group | Halt Medical Acessa Procedure
Number analyzed (Participants) | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 137
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years]
  Age US Sites (n=86) | 43.4 (4.0) [34 to 55]
  Age Latin America (n=51) | 40.7 (4.9) [31 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 86
  Mexico | 28
  Guatemala | 23

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Menstrual Blood Flow (MBF) at 12 Months Post Procedure
Description: Change in volume of menstrual blood loss at 12 months post-procedure compared to baseline. Bleeding relief and surgical reintervention were the co-primary endpoints. Bleeding relief success was defined for individual subjects as a ≥ 50% reduction from baseline in menstrual blood loss at 12 months posttreatment. The Primary Full Analysis Set was the primary analysis set for bleeding success rate.
Time Frame: 12 months from Baseline
Measure: Number; unit: Percentage of participants
Groups:
- Change of Menstrual Blood Flow(MBF) @ 12 Months Post Treatment: Of the 137 subjects enrolled and treated under this protocol, 124 (90.5%) were considered "evaluable" in terms of their 1) ability to provide a menstrual blood loss assessment, 2) lack of concomitant disease that affects the menstrual cycle, 3) baseline menstrual blood loss was within protocol inclusion limits.
Arm/Group | Change of Menstrual Blood Flow(MBF) @ 12 Months Post Treatment
Number analyzed (Participants) | 124
Percentage of participants
  50% change in MBF | 40.2 [31.6 to 48.7]
  40% change in MBF | 48.8 [40.1 to 57.5]
  30% change in MBF | 59.1 [50.5 to 67.6]
  22% change in MBF | 67.7 [59.6 to 75.8]

2. Primary Outcome: Incidence of Device and Procedure-related Adverse Events Within 12 Months Post-procedure
Description: An adverse event was defined as any untoward medical occurrence in a subject who uses a medical device, regardless of the presumed relationship of the event to the study device. A serious adverse event is defined as an untoward medical occurrence that results in death, is life threatening, requires or prolongs hospitalization, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect. Preexisting conditions (i.e., underlying diseases that were present before the adverse event reporting period began), re-intervention for failure to meet the study endpoints, and pregnancy were not reported as adverse events. All adverse events that occured during the study were recorded on the Adverse Event case report form (CRF). The investigator recorded the adverse event and assessed the relationship of the adverse event to the device and/or procedure; the coding of the events was reviewed by the Clinical Events Committee (CEC).
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Device Related Adverse Events: Device-related events are those that the investigator considered to be definitely, probably, or possibly related to the device.
- Procedural: Procedure-related events are those that the investigator considered to be definitely, probably, or possibly related to the procedure, including those related to abdominal entry and anesthesia.
Arm/Group | Device Related Adverse Events | Procedural
Number analyzed (Participants) | 137 | 137
participants | 5 | 33

3. Primary Outcome: Surgical Re-Intervention for Menorrhagia at 12 Months Post-treatment
Description: Patients who had surgical reintervention for bleeding prior to 12 months follow-up. Surgical reintervention success was defined as no surgical reintervention for menorrhagia within the 12-month posttreatment period.
Time Frame: 12 months from Baseline
Measure: Number; unit: participants
Groups:
- Surgical Reintervention 12 Months Post Treatment: The Per Protocol Set was the primary analysis set for surgical reintervention.
Arm/Group | Surgical Reintervention 12 Months Post Treatment
Number analyzed (Participants) | 124
participants | 0

4. Secondary Outcome: Change in Uterine and Fibroid Volume at 12 Months Post-procedure Compared to Pre-procedure (Baseline) as Measured With Contrast-enhanced MRI (Magnetic Resonance Imaging)
Description: Evaluate change from baseline in uterine volume and fibroid volume at 12 months post-procedure as measured by contrast-enhanced magnetic resonance imaging (MRI) measurements. Specifically, the outcomes of uterine and fibroid volume changes are expressed as a mean percentage of volume reduction. Treatment with RFA resulted in a reduction from baseline in total uterine and fibroid volume, as assessed by pretreatment and posttreatment MRI, at 3 and 12 months posttreatment.
Time Frame: 12 month from Baseline
Population: The Full Analysis Set (FAS) was used in the analysis of the change in total uterine and fibroid volumes between baseline and 12 months post treatment. Of the 137 Subjects enrolled, two were excluded from the FAS because they did not meet all of the inclusion/exclusion criteria.
Measure: Mean (95% Confidence Interval); unit: percentage of volume
Groups:
- Change in Uterine Volume: Uterine volume assessment 12 months post treatment via contrast enhanced MRI
- Change in Fibroid Volume: Fibroid volume assessment 12 months post treatment via contrast enhanced MRI
Arm/Group | Change in Uterine Volume | Change in Fibroid Volume
Number analyzed (Participants) | 128 | 119
percentage of volume | -25 (135.7) [-30.41 to -19.52] | -44.3 (47.98) [-50.84 to -37.84]

5. Secondary Outcome: Change in Fibroid Symptom Severity and Quality of Life Scores at 12 Months Post-procedure as Compared to Pre-procedure (Baseline) Using the Uterine Fibroid Symptom and Health Related Quality of Life (UFS-QoL) Assessment Tool.
Description: The Uterine Fibroid Symptom and Health Related Quality of Life (UFS-QoL) assessment tool measures symptom severity and Health related quality of life.
  Symptom Severity (SS) - high scores indicate greater symptoms (bad) and low scores indicate less symptoms (good). Scores range from 0 to 100. Since this outcome measure indicates "change" in symptoms, a negative number indicates a reduction in symptoms and therefore improvement.
  Health Related (HRQL) - high scores indicate better health state. Scores range from 0 to 100. Since this outcome measure indicates "change" in health and quality of life, a positive number indicates and improvement.
Time Frame: 12 months from Baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Full Analysis Set - Symptom Severity: All treated subjects who met all inclusion and exclusion criteria and who completed the Symptom Severity Questionnaire at Baseline and 12 months.
- Full Analysis Set - Health Related Quality of Life (HRQL): All treated subjects who met all inclusion and exclusion Criteria and who completed the HRQL questionnaire at both baseline and 12 months.
Arm/Group | Full Analysis Set - Symptom Severity | Full Analysis Set - Health Related Quality of Life (HRQL)
Number analyzed (Participants) | 129 | 129
Units on a scale | -34.93 (23.339) [10.2 to 48] | 42.12 (23.060) [33.5 to 42.9]

6. Secondary Outcome: Change in Score on Questionnaire - General Health Outcome at 12 Months Post-procedure as Compared to Pre-procedure Using the EQ-5D (a Standardized Instrument for Use as a Measure of Health Outcome)
Description: The EQ-5D is a standardized instrument with scores ranging from 0 to 100, for use as a measure of general health outcome, such as mobility, self-care, usual activities, pain/discomfort and anxiety and depression. An increase in the score post treatment indicates less disease burden.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Full Analysis Set - Month 12 Health Status Change: All subjects who completed the Health State Score Questionnaire (EQ-5D) at both baseline and at 12 months post treatment.
Arm/Group | Full Analysis Set - Month 12 Health Status Change
Number analyzed (Participants) | 128
Units on a scale | 15.2 (20.219) [71.7 to 99.9]

7. Secondary Outcome: Overall Subject Treatment Outcome and Satisfaction Using the Overall Treatment Evaluation (OTE)
Description: The Overall Treatment Evaluation Survey refers to whether the patient felt symptoms improved, worsened or remained the same post treatment.
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Groups:
- Overall, Satisfaction With Uterine Fibroid Treatment: Patients were asked, overall, how satisfied with their uterine fibroid treatment.
- How Effective Was This Treatment in Eliminating Symptoms: Patients were asked to respond in their opinion, how effective was this treatment in eliminating their symptoms.
Arm/Group | Overall, Satisfaction With Uterine Fibroid Treatment | How Effective Was This Treatment in Eliminating Symptoms
Number analyzed (Participants) | 124 | 124
percentage of patients
  Somewhat Satisfied/Effective | 12.1 | 14.5
  Moderately Satisfied/Effective | 21.0 | 29.8
  Very Satisfied/Effective | 61.3 | 50.0

ADVERSE EVENTS:
Time Frame: Baseline thru 36 months
Groups:
- Safety Set: The Safety Set consisted of all subjects treated in the study.
Arm/Group | Safety Set
Serious Adverse Events (participants affected / at risk) | 15/137
Other Adverse Events (participants affected / at risk) | 7/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=137)
Atelactasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Viral Infection with Otitis Media (Infections and infestations) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Uterine Hemorrhage (Reproductive system and breast disorders) | 1 (1)
Achilles tendon rupture and intervertebral disc repair (Musculoskeletal and connective tissue disorders) | 1 (1)
Laceration in serosa of colon (Surgical and medical procedures) | 1 (1)
Spontaneous Abortion (Reproductive system and breast disorders) | 1 (1)
Pelvic Abscess (Reproductive system and breast disorders) | 1 (1)
Hemiparesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
MVA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia, resulting in blood transfusion (Endocrine disorders) | 1 (2)
Pulmonary Embolus (Reproductive system and breast disorders) | 1 (1)
Mild Stroke (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=137)
Urinary Tract Infection (Infections and infestations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less